CLINICAL TRIAL: NCT01927003
Title: Direct and Reversed Dorsal Digito-metacarpal Flaps: A Review of 24 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBTS1308112; CHS130-00215 (Other: Hebei Clinical Trail Committee)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2010-04

CONDITIONS: Finger Injuries; Soft Tissue Injuries
Keywords: defect,; dorsal branch of the digital artery,; dorsal digital flap,; dorsal metacarpal artery flap.
MeSH Terms: conditions — Finger Injuries; Soft Tissue Injuries

ARMS (1):
- Surgical flap (Experimental): Dorsal digito-metacarpal flap is based on the dorsal digital artery and dorsal metacarpal artery.
  Interventions: Procedure: Dorsal digito-metacarpal flap

INTERVENTIONS:
Procedure: Dorsal digito-metacarpal flap — The dorsal digito-metacarpal flap is a vascular island flap based on the dorsal digital artery and dorsal metacarpal artery. It has a longer vascular pedicle and provides tissue coverage of similar quality as that of normal glabrous skin but not sacrifice the digital artery.

SUMMARY:
Multiple digital injuries are often complex and severe, and the commonly used local and regional flaps may not be feasible. The authors reconstruct soft tissue defects of the fingers using the dorsal digito-metacarpal flap and evaluate the efficacy of this technique.

DETAILED DESCRIPTION:
At final follow-up, we measure the sensibility of the flaps using the static 2-point discrimination test. The Static 2-point discrimination test determines the minimal distance at which a subject can sense the presence of two needle. The modified American Society for Surgery of the Hand guidalines are used to stratify discriminator measurements(excellent <6 mm, good 6-10 mm, fair 11-15 mm, poor >15 mm). Each area is tested 3 times with a Discriminator (Ali Med, Dedham, MA). Two out of 3 correct answers are considered proof of perception before proceeding to another lower value. We stopp at 4mm as a limit of 2PD and consider this normal. The measurements are performed at a single time point at final follow up.

ELIGIBILITY:
Inclusion Criteria:

* the injured and adjacent fingers are unable to be used as the donor due to multiple digital injuries
* a soft tissue defect > 1.5 cm in length with exposed bone or tendon
* the reverse DMA flap may not be appropriate for tissue reconstruction due to the concomitant injuries or due to the limitation of the rotation arc
* a patient between 15 and 60 years of age

Exclusion Criteria:

* concomitant injuries involved all the finger that precluded their use as donor sites
* a defect less than 1.5 cm in length
* injuries to the course of the vascular pedicle

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The Static 2-point discrimination test | 18 to 24months
  The Static 2-point discrimination test determines the minimal distance at which a subject can sense the presence of two needle. The modified American Society for Surgery of the Hand guidalines are used to stratify discriminator measurements(excellent <6 mm, good 6-10 mm, fair 11-15 mm, poor >15 mm). Each area is tested 3 times with a Discriminator (Ali Med, Dedham, MA). Two out of 3 correct answers are considered proof of perception before proceeding to another lower value. We stopped at 4mm as a limit of 2PD and considered this normal. The measurements are performed at a single time point at final follow up.

SECONDARY OUTCOMES:
Patient satisfaction | 18 to 24 months
  Patients report their satisfaction with the appearance of the flap and the donor site according to the Michigan Hand Outcomes Questionnaire that is based on a 5-point response scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Tangshan, Tangshan, Hebei, China

REFERENCES:
- [Result] Yang D, Morris SF. Reversed dorsal digital and metacarpal island flaps supplied by the dorsal cutaneous branches of the palmar digital artery. Ann Plast Surg. 2001 Apr;46(4):444-9. doi: 10.1097/00000637-200104000-00017. PMID 11324891
- [Derived] Chen C, Zhang W, Tang P. Direct and reversed dorsal digito-metacarpal flaps: a review of 24 cases. Injury. 2014 Apr;45(4):805-12. doi: 10.1016/j.injury.2013.11.002. Epub 2013 Nov 13. PMID 24315482